CLINICAL TRIAL: NCT04414397
Title: A Multicenter, Evaluator-blinded, Randomized, Parallel-group, Controlled Study of the Safety and Effectiveness of JUVÉDERM® VOLUMA® XC Injectable Gel for Correction of Temple Hollowing
Brief Title: A Study Evaluating JUVÉDERM® VOLUMA® XC Injectable Gel for Correction of Temple Hollowing in Adult Participants ≥ 22 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1878-702-008
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-03

CONDITIONS: Temple Hollowing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No Treatment then JUVÉDERM® VOLUMA® XC (Other): Participants received no treatment for 3 months during the Control Period. They either exited the study at Month 3 or received an optional treatment with JUVÉDERM® VOLUMA® XC injectable gel treatment in both temples during the Post-Control Period and an optional touch-up treatment 30 days later. Participants did not receive any treatment during the Maintenance Treatment Period.
  Interventions: Device: JUVÉDERM® VOLUMA® XC; Other: No-treatment control
- JUVÉDERM® VOLUMA® XC (Experimental): Participants received JUVÉDERM® VOLUMA® XC injectable gel treatment in both temples during the Control Period followed by an optional touch-up treatment 30 days later. Participants exited the study at Month 13 or received an optional maintenance treatment and were followed for 6 months during the Maintenance Treatment Period.
  Interventions: Device: JUVÉDERM® VOLUMA® XC

INTERVENTIONS:
Device: JUVÉDERM® VOLUMA® XC — JUVÉDERM® VOLUMA® XC injectable gel
Other: No-treatment control — Participants received no treatment for 3 months during the Control Period.
  Arms: No Treatment then JUVÉDERM® VOLUMA® XC

SUMMARY:
The objectives of this study are to evaluate the safety and effectiveness of Juvederm® Voluma® XC injectable gel in adult participants seeking correction of temple hollowing

ELIGIBILITY:
Inclusion Criteria:

* Participants in general good health
* Participants seeking improvement of temple hollowing

Exclusion Criteria:

* Temple hollowing due to trauma, congenital malformations, or lipodystrophy
* Temporomandibular joint dysfunction or any other jaw issues
* Recurrent temporal headaches such as temporal tendinitis migraine
* Active autoimmune disease
* History of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), HA products, or Streptococcal protein
* Prior facial reconstructive surgeries, facelift, or browlift as well as surgeries on the temple area (eg, biopsy)
* Fat injection or permanent facial implants anywhere in the face
* Semipermanent soft-tissue filler treatment in the temple or mid-face within 36 months before enrollment
* Temporary dermal filler injections above the subnasale within 24 months before enrollment
* Mesotherapy or cosmetic facial procedures above the subnasale within 6 months before enrollment
* Botulinum toxin treatment above the subnasale within 6 months before enrollment
* Females who are pregnant, nursing, or planning a pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN, INC., Study Director — Allergan
Locations (15):
- United States (14):
  - Skin Care and Laser Physicians of Beverly Hills /ID# 232967, Los Angeles, California
  - Steve Yoelin MD Medical Associate Inc /ID# 232956, Newport Beach, California
  - Steven Fagien MD PA /ID# 232807, Boca Raton, Florida
  - Bradenton Dermatologist /ID# 232822, Bradenton, Florida
  - Hevia Cosmetic Dermatology /ID# 232824, Coral Gables, Florida
  - Skin and Cancer Associates, LLP /ID# 232923, Miami, Florida
  - Research Institute of the Southeast, LLC /ID# 233144, West Palm Beach, Florida
  - Delricht Research /ID# 233142, New Orleans, Louisiana
  - Callender Center for Clinical Research /ID# 233167, Glenn Dale, Maryland
  - Skincare Physicians /ID# 233054, Chestnut Hill, Massachusetts
  - Williams Plastic Surgery Specialists /ID# 232789, Latham, New York
  - Aesthetic Solutions /ID# 232953, Chapel Hill, North Carolina
  - The Practice of Brian S. Biesman MD PLLC /ID# 232662, Nashville, Tennessee
  - Dallas Plastic Surgery Institute /ID# 232971, Dallas, Texas
- Jose Raul Montes Eyes & Facial Rejuvenation-Torre Medica Aux /ID# 232706, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=1878-702-008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 205 participants screened, 171 were randomized, with 113 in the treatment group and 58 in the control group. One participant was randomized to the treatment group but not treated.
Period: Control Period
Arm/Group | No Treatment Then JUVÉDERM® VOLUMA® XC | JUVÉDERM® VOLUMA® XC
Started | 58 | 113 (One participant was randomized but not treated.)
Completed | 56 | 106
Not Completed | 2 | 7
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 4
Not completed — Protocol deviation | 0 | 1
Period: Post-Control Period
Arm/Group | No Treatment Then JUVÉDERM® VOLUMA® XC | JUVÉDERM® VOLUMA® XC
Started | 53 | 106
Completed | 46 | 91
Not Completed | 7 | 15
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lost to Follow-up | 4 | 9
Period: Maintenance Treatment Period
Arm/Group | No Treatment Then JUVÉDERM® VOLUMA® XC | JUVÉDERM® VOLUMA® XC
Started | 0 | 40
Completed | 0 | 35
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat Population(mITT): all participants who were randomized and had non-missing Baseline Allergan Temple Hollowing Scale (ATHS) scores. Participants were summarized according to the randomized study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment Then JUVÉDERM® VOLUMA® XC | JUVÉDERM® VOLUMA® XC | Total
Number analyzed (Participants) | 58 | 113 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (9.81) | 54.9 (9.97) | 54.7 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 96 | 143
  Male | 11 | 17 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 27 | 41
  Not Hispanic or Latino | 44 | 86 | 130
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 12 | 18
  White | 48 | 94 | 142
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 1-grade Improvement From Baseline in the Validated Allergan Temple Hollowing Scale (ATHS) Based on Evaluating Investigator (EI) Assessment at Month 3
Description: The Evaluating Investigator assessed the participant's temple hollowing using the 5-point ATHS scale where 0=convex, rounded temple and 4=severe, deeply recessed, sunken appearance. A 1-point decrease from Baseline indicates improvement.
Time Frame: Baseline, Month 3 (Control Period)
Population: Modified Intent to Treat Population(mITT): all participants who were randomized and had non-missing Baseline Allergan Temple Hollowing Scale (ATHS) scores. Participants were summarized according to the randomized study intervention. Multiple imputation was used for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No Treatment Then JUVÉDERM® VOLUMA® XC | JUVÉDERM® VOLUMA® XC
Number analyzed (Participants) | 58 | 113
percentage of participants | 13.5 [4.5 to 22.5] | 80.4 [72.7 to 88.1]
Statistical Analysis 1: Comparison: No Treatment Then JUVÉDERM® VOLUMA® XC vs JUVÉDERM® VOLUMA® XC; JUVÉDERM® VOLUMA® XC Treatment vs No-treatment control; Test type: Superiority; p < 0.0001, Multiple imputation regression — Analysis was performed using the SAS procedure MIANALYZE with normal approximation to generate an associated p-value for the comparison of responder rates between groups; Rate Difference = 66.9, 95% CI 2-sided [54.9 to 78.8]

2. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant whether or not it is related to the investigational product. The investigator assesses the relationship of each event to the use of the investigational product. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first use of the investigational product.
Time Frame: From the time of informed consent until the participant exited the study, up to 13 months after their initial/touch-up treatment, and up to 6 months after the maintenance treatment
Population: Safety population: all participants who were randomized and received study intervention (JUVÉDERM® VOLUMA® XC or no-treatment control), analyzed by treatment received
Measure: Count of Participants; unit: Participants
Groups:
- No Treatment (Control Period): Participants who received no treatment during the first 3 months of the Control Period.
- JUVÉDERM® VOLUMA® XC (Control Period + Post-Control Period): Participants received JUVÉDERM® VOLUMA® XC injectable gel treatment in both temples during the Control Period followed by an optional touch-up treatment 30 days later. They were followed up to Month 13.
- JUVÉDERM® VOLUMA® XC (Post-Control Period): Participants received an optional treatment with JUVÉDERM® VOLUMA® XC injectable gel treatment in both temples during the Post-Control Period and an optional touch-up treatment 30 days later. They were followed up to Month 13.
- JUVÉDERM® VOLUMA® XC (Maintenance Period): Participants received an optional maintenance treatment and were followed for 6 months during the Maintenance Treatment Period.
Arm/Group | No Treatment (Control Period) | JUVÉDERM® VOLUMA® XC (Control Period + Post-Control Period) | JUVÉDERM® VOLUMA® XC (Post-Control Period) | JUVÉDERM® VOLUMA® XC (Maintenance Period)
Number analyzed (Participants) | 59 | 112 | 53 | 40
Participants
  Any TEAE | 3 | 38 | 24 | 13
  TESAE | 2 | 5 | 2 | 4

3. Secondary Outcome: Percentage of Participants With a Score of "Improved " or "Much Improved" on the Global Aesthetic Improvement Scale (GAIS) for the Temple Area as Assessed by the Evaluating Investigator (EI) at Month 3
Description: The Evaluating Investigator assessed the participant's temple area using the 5-point GAIS where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse.
Time Frame: Month 3 (Control Period)
Population: Modified Intent to Treat Population(mITT): all participants who were randomized and had non-missing Baseline Allergan Temple Hollowing Scale (ATHS) scores. Participants were summarized according to the randomized study intervention. Participants with analysis values at Month 3 are presented.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No Treatment Then JUVÉDERM® VOLUMA® XC | JUVÉDERM® VOLUMA® XC
Number analyzed (Participants) | 56 | 105
percentage of participants | 10.7 [4.0 to 21.9] | 83.8 [75.3 to 90.3]

4. Secondary Outcome: Percentage of Participants With a Score of "Improved" or "Much Improved" on the Global Aesthetic Improvement Scale (GAIS) for the Temple Area as Assessed by the Participants at Month 3
Description: Participants assessed their temple area using the 5-point GAIS where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse.
Time Frame: Month 3 (Control Period)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No Treatment Then JUVÉDERM® VOLUMA® XC | JUVÉDERM® VOLUMA® XC
Number analyzed (Participants) | 51 | 99
percentage of participants | 2.0 [0.0 to 10.4] | 92.9 [86.0 to 97.1]

5. Secondary Outcome: Change From Baseline on FACE-Q Satisfaction With Facial Appearance Questionnaire at Month 3
Description: The participants responded to each item on the FACE-Q Satisfaction with Facial Appearance questionnaire using a 4-point scale where: 1=Very Dissatisfied, 2=Somewhat Dissatisfied, 3=Somewhat Satisfied, and 4=Very Satisfied. The total score was transformed to a score of 0 (worst) to 100 (best) for comparison. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 3 (Control Period)
Population: Modified Intent to Treat Population(mITT): all participants who were randomized and had non-missing Baseline Allergan Temple Hollowing Scale (ATHS) scores. Participants were summarized according to the randomized study intervention. Overall number of participants analyzed were the participants with analysis values at both Baseline and Month 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Treatment Then JUVÉDERM® VOLUMA® XC | JUVÉDERM® VOLUMA® XC
Number analyzed (Participants) | 51 | 100
units on a scale | -6.6 (8.90) | 24.2 (22.32)
Statistical Analysis 1: Comparison: JUVÉDERM® VOLUMA® XC; Test type: Other; p < 0.0001, t-test, 2 sided — P-value is based on a 2-sided paired t-test at the 5% level to demonstrate that the mean satisfaction score at Month 3 visit is statistically greater than at Baseline for the treatment group

6. Secondary Outcome: Change From Baseline to Month 3 on Participants Responses on FACE-Q Satisfaction With Temples Questionnaire
Description: The participants responded to each item on the FACE-Q Satisfaction with Temples questionnaire using a 4-point scale where: 1=Very Dissatisfied, 2=Somewhat Dissatisfied, 3=Somewhat Satisfied, 4=Very Satisfied. The total score was transformed to a score of 0 (worst) to 100 (best) for comparison. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Month 3 (Control Period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Treatment Then JUVÉDERM® VOLUMA® XC | JUVÉDERM® VOLUMA® XC
Number analyzed (Participants) | 51 | 100
units on a scale | -4.2 (14.77) | 42.7 (26.65)
Statistical Analysis 1: Comparison: JUVÉDERM® VOLUMA® XC; Test type: Other; p < 0.0001, t-test, 2 sided — P-value is based on a 2-sided paired t-test at the 5% level to demonstrate that the mean satisfaction score at Month 3 is statistically greater than at Baseline for the treatment group

ADVERSE EVENTS:
Time Frame: No Treatment (Control Period): from the time of consent up to Month 3 JUVÉDERM® VOLUMA® XC (Control Period + Post-Control Period): from the time of consent up to Month 13 JUVÉDERM® VOLUMA® XC (Post-Control Period): from the time of treatment up to Month 13 JUVÉDERM® VOLUMA® XC (Maintenance Period): from the time of maintenance treatment up to Month 6
Description: Safety population: all participants who were randomized and received study intervention, analyzed by treatment received
Groups:
- JUVÉDERM® VOLUMA® XC (Post-Control Period): Participants randomized to no treatment during the first 3 months of the Control Period who then received an optional treatment with JUVÉDERM® VOLUMA® XC injectable gel treatment in both temples during the Post-Control Period and an optional touch-up treatment 30 days later. They were followed up to Month 13.
- JUVÉDERM® VOLUMA® XC (Maintenance Period): Participants randomized to JUVÉDERM® VOLUMA® XC injectable gel treatment in both temples during the Control Period who then received an optional maintenance treatment and were followed for 6 months during the Maintenance Treatment Period.
Arm/Group | No Treatment (Control Period) | JUVÉDERM® VOLUMA® XC (Control Period + Post-Control Period) | JUVÉDERM® VOLUMA® XC (Post-Control Period) | JUVÉDERM® VOLUMA® XC (Maintenance Period)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/112 | 0/53 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/59 | 5/112 | 2/53 | 4/40
Other Adverse Events (participants affected / at risk) | 0/59 | 19/112 | 16/53 | 5/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Treatment (Control Period) (N=59) | JUVÉDERM® VOLUMA® XC (Control Period + Post-Control Period) (N=112) | JUVÉDERM® VOLUMA® XC (Post-Control Period) (N=53) | JUVÉDERM® VOLUMA® XC (Maintenance Period) (N=40)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYME DISEASE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Treatment (Control Period) (N=59) | JUVÉDERM® VOLUMA® XC (Control Period + Post-Control Period) (N=112) | JUVÉDERM® VOLUMA® XC (Post-Control Period) (N=53) | JUVÉDERM® VOLUMA® XC (Maintenance Period) (N=40)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (11) | 7 (9) | 1 (2)
TRISMUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (3) | 2 (3)
HEADACHE (Nervous system disorders) | 0 (0) | 9 (10) | 9 (10) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT04414397/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT04414397/SAP_001.pdf